CLINICAL TRIAL: NCT06058052
Title: Pattern Of Association Between Obstructive Seep Apnea and Interstitial Lung Disease
Brief Title: Prevalence of OSA in Patients of ILD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Doctor, Assiut University
Other Study IDs: ILD,OSA
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-04

CONDITIONS: OSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the clinical predictors of OSA in patients with ILD

DETAILED DESCRIPTION:
Interstitial lung diseases (ILDs) are a group of heterogeneous disorders characterized by varying degrees of fibrosis and inflammation of lung parenchyma.

Obstructive sleep apnea is a type of sleep disordered breathing characterized by repeated episodes of apnea and hypopnea during sleep due to narrowing or occlusion of the upper airway.

It was found that the prevalence of OSA is as high as 80% among patients with idiopathic pulmonary fibrosis (IPF). Despite this common association, there is limited research in this field. There is great need for further studies to highlight this association and understand the underlying pathophysiological mechanisms implicated in those patients, to ultimately guide the appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to Chest Department with interstitial lung disease will be included, screened for OSA.

Exclusion Criteria:

* Age: less than 18 years. Unstable patients or need for ICU admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Assiut University Hospital diagnosed as interstitial lung disease risky for OSA will be included from June 2023 to January 2024.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-09-28 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Predictors of OSA in patients with ILD | Baseline
  By clinical history ,examination, BMI

SECONDARY OUTCOMES:
Prevalence of OSA among patients with ILD Presented To Chest Department in Assiut University Hospital | base line
  BY Polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed yassen, MD, Study Chair — Assiut University